CLINICAL TRIAL: NCT01331993
Title: A Phase I, Open-label, Randomised, 3-way Crossover Study to Demonstrate Bioequivalence of a Single Oral Dose of Naproxen Administered as VIMOVO Manufactured at AstraZeneca AB Compared to That of VIMOVO Manufactured by Patheon Pharmaceuticals and a Marketed Enteric-coated Naproxen Formulation (Manufactured by Roche) in Healthy Volunteers
Brief Title: A Bioequivalence Study to Compare VIMOVO Manufactured at AstraZenca AB to VIMOVO Manufactured by Patheon Pharmaceuticals and Marketed Enteric-coated Naproxen Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1120C00030
Record Dates: First submitted 2011-03-11; First posted 2011-04-08 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteers; Bioequivalence
Keywords: Phase 1; crossover; bioequivalence; naproxen; esomeprazole; vimovo; healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Treatment order : A, B, C
  Interventions: Drug: VIMOVO (AstraZeneca); Drug: VIMOVO (Patheon); Drug: Marketed enteric-coated naproxen formulation
- 2 (Experimental): Treatment order : B, C, A
  Interventions: Drug: VIMOVO (AstraZeneca); Drug: VIMOVO (Patheon); Drug: Marketed enteric-coated naproxen formulation
- 3 (Experimental): Treatment order : C, A, B
  Interventions: Drug: VIMOVO (AstraZeneca); Drug: VIMOVO (Patheon); Drug: Marketed enteric-coated naproxen formulation
- 4 (Experimental): Treatment order : A, C, B
  Interventions: Drug: VIMOVO (AstraZeneca); Drug: VIMOVO (Patheon); Drug: Marketed enteric-coated naproxen formulation
- 5 (Experimental): Treatment order : B, A, C
  Interventions: Drug: VIMOVO (AstraZeneca); Drug: VIMOVO (Patheon); Drug: Marketed enteric-coated naproxen formulation
- 6 (Experimental): Treatment order : C, B, A
  Interventions: Drug: VIMOVO (AstraZeneca); Drug: VIMOVO (Patheon); Drug: Marketed enteric-coated naproxen formulation

INTERVENTIONS:
Drug: VIMOVO (AstraZeneca) — VIMOVO (AstraZeneca) 500 mg naproxen/20 mg esomeprazole
  Other Names: Treatment A
Drug: VIMOVO (Patheon) — VIMOVO (Patheon) 500 mg naproxen/20 mg esomeprazole
  Other Names: Treatment B
Drug: Marketed enteric-coated naproxen formulation — Marketed enteric-coated naproxen formulation (manufactured by Roche) 500 mg tablet
  Other Names: Treatment C

SUMMARY:
The primary purpose is to demonstrate the bioequivalence of naproxen administered as VIMOVO manufactured at a new facility in Sweden (AstraZeneca) to that of naproxen administered as VIMOVO manufactured in the USA (Patheon) and to a marketed enteric-coated naproxen formulation.

DETAILED DESCRIPTION:
A Phase I, Open-label, Randomised, 3-way Crossover Study to demonstrate Bioequivalence of a Single Oral Dose of Naproxen administered as VIMOVO manufactured at AstraZeneca AB compared to that of VIMOVO manufactured by Patheon Pharmaceuticals and a marketed enteric-coated Naproxen Formulation (Manufactured by Roche) in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteer, aged 18 - 55 years (inclusive)
* Female volunteers must be non-pregnant and non-lactating and have a negative urine pregnancy test result prior to enrolment into the study.
* Female volunteers of childbearing potential must be using appropriate birth control during the entire duration of the study
* Body mass index of = 19 to =30 kg/m2 (inclusive) and weights of = 50 to = 100 kg (inclusive)

Exclusion Criteria:

* Volunteer who is likely to have unrecognized cardiovascular or cerebrovascular disease, based on history or risk factors, or who has a clinical significant ECG finding at screening
* Uncontrolled hypertension defined as resting systolic pressure >140 mmHg or diastolic pressure >90 mmHg at screening or admission to Period 1
* Presence or prior history of abnormal bleeding or bleeding disorders, or any volunteer with significant history of peptic ulcer disease or other acid related gastrointestinal symptoms
* Any gastrointestinal disease, abnormality or gastric surgery that may interfere with gastric emptying, motility and drug absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in area under the plasma concentration-time curve (AUC) from time zero to infinity | Pre-dose to Day 4

SECONDARY OUTCOMES:
Number of subjects with Adverse Events as a measure of Safety and Tolerability | Day 1
Number of subjects with Adverse Events as a measure of Safety and Tolerability | Day 2
Number of subjects with Adverse Events as a measure of Safety and Tolerability | Day 3
Number of subjects with Adverse Events as a measure of Safety and Tolerability | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Stepehn Kanes, Study Director — AstraZeneca, Wilmington, USA; Kingsley Urakpo, MD, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital, 6 Newcomen St, London SE1 1YR, UK
Locations (1):
- Research Site, London, United Kingdom